CLINICAL TRIAL: NCT00992342
Title: A Double Blind (3rd Party Open), Randomised, Placebo-Controlled, Dose Escalation Study To Investigate The Safety, Toleration, And Pharmacokinetics Of Multiple Oral Doses Of PF-03893787 In Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate The Safety And Tolerability Of Different Doses Of PF-03893787 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0281003
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-03893787 5 mg (Experimental)
  Interventions: Drug: PF-03893787
- PF-03893787 15 mg (Experimental)
  Interventions: Drug: PF-03893787
- PF-03893787 50 mg (Experimental)
  Interventions: Drug: PF-03893787

INTERVENTIONS:
Drug: PF-03893787 — oral solution, 5 mg, QD for 14 days
  Arms: PF-03893787 5 mg
Drug: PF-03893787 — oral solution, 15 mg, QD for 14 days
  Arms: PF-03893787 15 mg
Drug: PF-03893787 — oral solution, 50 mg, QD for 14 days
  Arms: PF-03893787 50 mg

SUMMARY:
The purpose of this study is to investigate safety and toleration of multiple oral doses as well as the time course of PF-03893787 concentration in the blood following dosing by oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and females of non-childbearing potential between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males and 14 drinks/week for females.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety/toleration: Adverse events, vital signs, 12 lead ECG, blood (including creatine kinase) and urine safety tests and physical examination. | 22 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Cmax, Tmax, AUCτ, t½, accumulation ratio, | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0281003&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20Different%20Doses%20Of%20PF-03893787%20In%20Healthy%20Adult%20Volunteers